CLINICAL TRIAL: NCT03985358
Title: A Prospective Randomized Study Analyzing Preoperative Opioid Counseling in Pain Management After Reduction Mammoplasty
Brief Title: Opioid Counseling in Pain Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00037881
Record Dates: First submitted 2018-10-25; First posted 2019-06-13 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Pain, Postoperative
Keywords: opioid counseling; bilateral reduction mammoplasty
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Randomized, controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Patients randomized to the Control Group will not receive opioid counseling and will only receive their standard of care instructions for preoperative and postoperative care.
- Treatment Group (Experimental): Patients randomized to the Treatment Group will have opioid counseling plus standard of care instructions given by the same counselor (investigator on the study) using the same counseling script at the randomization visit as well as at the visit where they come in for pre-admission testing prior to surgery (as a refresher).
  Interventions: Other: Opioid counseling plus standard of care instructions

INTERVENTIONS:
Other: Opioid counseling plus standard of care instructions — Same counselor (investigator on the study) will use the same counseling script at the randomization visit as well as at the visit where they come in for pre-admission testing prior to surgery (as a refresher) to counsel patients
  Arms: Treatment Group

SUMMARY:
The purpose of this study is to evaluate the effect of perioperative opioid counseling within a specific group of patient population who are undergoing bilateral reduction mammoplasty.

DETAILED DESCRIPTION:
Prescription opioid abuse has been increasing dramatically in recent years. There is growing concern regarding the unprecedented increase in morbidity and mortality related to the use of opioids.1-2 In 2010 the rates of opioid sales, deaths, as well as associated treatment admissions have increased to more than triple the rates in 1999.1-2 Although policy makers and the media often associate the opioid crisis as a problem of nonmedical opioid abuse, evidence has suggested that opioid addiction occurs in both medical and nonmedical users.2 The Centers for Disease control and Prevention reported and warned that long-term opioid use often starts with treatment of some type of acute pain.3 Prescription opioids have been shown to be favorable in perioperative pain management, however, their effectiveness in chronic pain management is not as clear. Surgeons are among the highest opioid prescribers. Many common elective as well as trauma-related procedures have been reported as possible causes of increased prolonged opioid usage. Recent evidence also suggested that a considerable number of patients who were prescribed opioids struggle to with transitioning to non-opioid pain medications.1-6 Numerous methods have been considered and explored in effort of decreasing the misuse and abuse of prescription opioids. One of the methods being opioid counseling, in which patients are educated on the effects and risks of short-term and long-term opioid usage and physicians recommend and discuss the appropriate opioid usage as well as alternative nonopioid options. It has also been indicated that counseling is more effective if given earlier on in the patient's surgical care rather than through rushed education overview at discharge.1,4-6 Therefore, the purpose of this study is to evaluate the effect of perioperative opioid counseling within a specific group of patient population who are undergoing bilateral reduction mammoplasty.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Elective bilateral reduction mammoplasty to be performed as outpatient
* Able and willing to provide informed consent
* Able and willing to comply with study procedures

Exclusion Criteria:

* Age < 18 years
* Bilateral reduction mammoplasty planned/performed with any concomitant procedures
* History of preoperative opioid consumption or rehabilitation
* Opioid allergy
* Local anesthetic given during or after procedure
* Unable and/or unwilling to provide informed consent
* Unable and/or unwilling to comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Pain level | 1 month
  using standard pain scale scores recorded in daily diary - using scale 0 to 10 with 0 being "no pain" and 10 being "worst pain imaginable"
Opioid consumption | 1 month
  pain pill counts
Patient satisfaction | 3 months
  Satisfied versus not satisfied with pain management using rating categories of: very satisfied, satisfied, neutral, dissatisfied, and very dissatisfied

CONTACTS AND LOCATIONS:
Overall Officials: Wilton Triggs, MD, Principal Investigator — University of South Florida
Locations (1):
- Tampa General Hospital, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim N, Matzon JL, Abboudi J, Jones C, Kirkpatrick W, Leinberry CF, Liss FE, Lutsky KF, Wang ML, Maltenfort M, Ilyas AM. A Prospective Evaluation of Opioid Utilization After Upper-Extremity Surgical Procedures: Identifying Consumption Patterns and Determining Prescribing Guidelines. J Bone Joint Surg Am. 2016 Oct 19;98(20):e89. doi: 10.2106/JBJS.15.00614. PMID 27869630
- [Background] Costello M. Prescription Opioid Analgesics: Promoting Patient Safety with Better Patient Education. Am J Nurs. 2015 Nov;115(11):50-6. doi: 10.1097/01.NAJ.0000473315.02325.b4. PMID 26510070
- [Background] Holman JE, Stoddard GJ, Horwitz DS, Higgins TF. The effect of preoperative counseling on duration of postoperative opiate use in orthopaedic trauma surgery: a surgeon-based comparative cohort study. J Orthop Trauma. 2014 Sep;28(9):502-6. doi: 10.1097/BOT.0000000000000085. PMID 24667804
- [Result] Alter TH, Ilyas AM. A Prospective Randomized Study Analyzing Preoperative Opioid Counseling in Pain Management After Carpal Tunnel Release Surgery. J Hand Surg Am. 2017 Oct;42(10):810-815. doi: 10.1016/j.jhsa.2017.07.003. Epub 2017 Sep 8. PMID 28890331
- [Result] Kolodny A, Courtwright DT, Hwang CS, Kreiner P, Eadie JL, Clark TW, Alexander GC. The prescription opioid and heroin crisis: a public health approach to an epidemic of addiction. Annu Rev Public Health. 2015 Mar 18;36:559-74. doi: 10.1146/annurev-publhealth-031914-122957. Epub 2015 Jan 12. PMID 25581144
- [Result] Johnson SP, Chung KC, Zhong L, Shauver MJ, Engelsbe MJ, Brummett C, Waljee JF. Risk of Prolonged Opioid Use Among Opioid-Naive Patients Following Common Hand Surgery Procedures. J Hand Surg Am. 2016 Oct;41(10):947-957.e3. doi: 10.1016/j.jhsa.2016.07.113. Epub 2016 Sep 28. PMID 27692801